CLINICAL TRIAL: NCT06954441
Title: V-IMMUNE® for Primary Immunodeficiency: A Phase III Clinical Trial (VIP Study)
Brief Title: V-IMMUNE: A Novel Immunoglobulin Therapy for Immunodeficiency
Acronym: VIP
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: On Pharma Importadora, Exportadora e Distribuidora de Medicamentos LTDA. (Other)
Collaborators: Hospital do Coracao (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VIP study
Record Dates: First submitted 2025-04-15; First posted 2025-05-01 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-04

CONDITIONS: Immunodeficiencies; Primary Immunodeficiencies (PID); Agammaglobulinemia
Keywords: immunodeficiency; intravenous immunoglobulin; pharmacokinetics; safety; efficacy; serious bacterial infection; temporally related adverse event
MeSH Terms: conditions — Immunologic Deficiency Syndromes; Agammaglobulinemia | interventions — Immunoglobulins, Intravenous; V-Set Domain-Containing T-Cell Activation Inhibitor 1

STUDY DESIGN:
Intervention Model Description: All participants will get the same intervention: IV immunoglobulin each 3 weeks. Participants meeting the inclusion criteria will receive V-IMMUNE® at a dose of 600 mg/kg, with infusion rates progressively increased to a maximum of 0.06 mL/kg/min, provided no adverse events occur. Pre-medication with intravenous normal saline, hydrocortisone and diphenhydramine is administered to mitigate infusion-related risks.
Masking Description: no masking
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention arm (Experimental): Human normal immunoglobulin I.P. 5% (5 g/100 mL) V-IMMUNE® will be administered at a dose of 600 mg/kg every 3 weeks (±3 days) via intravenous (IV) infusion according to the rate below, over a duration of 3 to 6 hours (4):
  0.01 mL/kg/min from 0 to 30 minutes, followed by the following infusion rates: 0.02 mL/kg/min from 31 to 45 minutes 0.04 mL/kg/min from 46 to 60 minutes 0.06 mL/kg/min from 61 minutes until the end of the infusion The dose increases gradually unless adverse events (AEs) occur. The infusion rate is only increased if the patient tolerates it well, with no AEs.
  If an AE occurs, the infusion must be interrupted for 20 to 30 minutes. Pre-medication: 30 to 60 min before Ig Rapid administration of 500 mL of 0.9% NaCl IV Diphenhydramine* 50 mg IV (adult). Pediatrics: 1.25 mg/kg IV Hydrocortisone** 200 mg IV (adult). Pediatrics: 3 mg/kg IV After infusion: 0.9% NaCl at 1 mL/kg/hour for one hour After three months, diphenhydramine and hydrocortisone may no loger be needed
  Interventions: Biological: Intravenous immunoglobulin (IVIG)

INTERVENTIONS:
Biological: Intravenous immunoglobulin (IVIG) — The investigational product is V-IMMUNE®, a 5% human normal immunoglobulin I.P. (5 g/100 mL) manufactured from qualified human plasma for intravenous use. Each vial contains human immunoglobulin at 50 g/L, maltose at 100 g/L, and water for injection. The 5% Human Immunoglobulin Solution for Intravenous Administration (I.P.) is a sterile and pyrogen-free preparation of human normal immunoglobulin in a single-dose form for intravenous administration. Each 10 mL, 50 mL, or 100 mL vial contains 0.5 g, 2.5 g, or 5 g of human normal immunoglobulin, respectively, and is produced from qualified human plasma using membrane filtration and a combination of chromatographic steps and viral inactivation procedures. The IgA content does not exceed 2 mg/mL.
  This manufacturing process uses plasma collected from donors who undergo screening according to guidelines set by regulatory authorities.
  In case of thromboembolic risk: use the lowest feasible dose
  Other Names: V-IMMUNE

SUMMARY:
This is a phase III, non-randomized clinical trial (VIP Study) designed to assess the safety and efficacy of V-IMMUNE®, a 5% human normal immunoglobulin preparation, in approximately 50 patients with primary immunodeficiency (PID). Participants, all aged ≥2 years and already receiving IVIG therapy, will be switched to V-IMMUNE® at a dose of 600 mg/kg every three weeks via intravenous infusion. The study will use historical data as a control and extend over 12 months, with scheduled visits at each infusion (an estimated 17 infusions per participant).

Objectives and Outcomes Primary Efficacy Endpoint: Rate of serious bacterial infections over 12 months. Primary Safety Endpoint: Proportion of infusions with one or more temporally associated adverse events (AEs).

Secondary Endpoints: Additional safety outcomes (e.g., average number of AEs within 72 hours per infusion), efficacy measures (non-serious bacterial infections, time to resolution, antibiotic use, hospitalizations), and quality of life (SF-36) at 6 and 12 months. A pharmacokinetic (PK) sub-study will be conducted in 20 participants aged ≥16 years to evaluate total IgG levels, half-life, AUC, Cmax, and other PK parameters.

Study Design and Intervention V-IMMUNE® is given at an initial infusion rate of 0.01 mL/kg/min for 30 minutes, increasing stepwise up to 0.06 mL/kg/min if well tolerated. Pre-medication, including rapid IV saline, diphenhydramine, and hydrocortisone, will be administered for the first three months to reduce the risk of infusion-related AEs. Patients at elevated thromboembolic risk will receive the lowest feasible infusion rate.

Sample Size and Analysis Fifty patients total will be enrolled to ensure adequate power to demonstrate a severe infection rate below one event per person-year (with a one-sided 1% significance level). Safety endpoints will be met if the upper bound of the 95% confidence interval for the proportion of temporally associated infusion-related AEs remains below 40%, assuming a true rate under 20%. An interim analysis is planned at six months or upon reaching 50% enrollment.

20 patients at total including adults and <16 years old, 6 children from 2 to 12 years old and 6 children from 12 to 16 years old.

DETAILED DESCRIPTION:
Introduction:

Immunoglobulin is used as a treatment for a variety of medical conditions, not only for its ability to combat infection as replacement therapy, but also for its anti-inflammatory and immunomodulatory effects. Immunoglobulins are primarily characterized by their antibody function, with various classes and subclasses that perform different roles. B cells are primarily responsible for the humoral adaptive immune response (antibody-mediated). Immunoglobulins, which are the molecules with antibody function, serve as the receptors of B cells, anchored to the membrane via a molecular complex composed of molecules that both anchor the immunoglobulin and promote signal transduction into the cell. This enables B cell activation, triggering a signaling cascade that leads to terminal differentiation into plasma cells or memory cells.

Inborn errors of immunity (primary immunodeficiencies - PIDs) represent a large, heterogeneous, and rapidly growing group of genetic diseases, primarily (but not exclusively) caused by loss- or gain-of-function germline mutations in genes associated with the immune response. Despite their individual rarity, inborn errors collectively affect a significant proportion of patients, with an estimated global prevalence of 1 in 1,200-2,000. They now comprise approximately 500 known genetic causes, subdivided into 10 categories listed in the 2022 classification by the International Union of Immunological Societies (IUIS), about two-thirds of which have been identified in the past decade. As evidence of the field's dynamic development, approximately 30 new diseases have been described per year in recent years.

Worldwide, the most common defects among PIDs-approximately 60%-involve impaired antibody production, with selective IgA deficiency and common variable immunodeficiency being the most prevalent. At least 80% of patients diagnosed with antibody deficiency receive IgG replacement therapy. PIDs can be an unrecognized underlying condition associated with autoimmune, allergic, and lymphoproliferative diseases and may therefore remain undiagnosed for many years. Patients diagnosed with B cell dysfunction and resulting antibody deficiencies require immunoglobulin G (IgG) replacement, a safe and effective therapeutic option for preventing infections in patients with PIDs.

Intravenous immunoglobin is used to treat a wide range of diseases. However, its approved indications can be divided into three main categories: primary and secondary antibody deficiencies, vertically transmitted HIV, chronic lymphocytic leukemia (CLL), immune thrombocytopenic purpura (ITP), chronic inflammatory demyelinating polyneuropathy (CIDP), severe disseminated infections, and graft-versus-host disease. It is recommended to initiate immunoglobulin replacement therapy in all patients who meet the diagnostic criteria for IgG hypogammaglobulinemia, whether they have agammaglobulinemia, common variable immunodeficiency (CVID), or IgG subclass deficiencies with functional antibody production impairment In this protocol, investigators discuss the use of a commercially available human polyvalent immunoglobulin product for intravenous use at 5% concentration, branded V-MMUNE, for the treatment of inborn errors of humoral immunity / primary immunodeficiencies involving impaired production of IgG class immunoglobulins by B lymphocytes.

Considering the relative unavailability of blood products, among which immunoglobulins are in the most critical category, the approval of new products in Brazil is of utmost importance due to the increasing need for this medication-even for well-defined indications such as hypogammaglobulinemia, whether primary or secondary, as well as neuropathies like Guillain-Barré syndrome, chronic inflammatory demyelinating polyneuropathy (CIDP), and hematologic conditions such as immune thrombocytopenic purpura. Several factors have contributed to this shortage, including increasingly stringent safety requirements; the difficulty in obtaining high-quality plasma that meets the standards of major regulatory agencies such as the FDA and EMA; the need to improve manufacturing processes; the reduction in the number of donors due to the COVID-19 pandemic; and the increased demand for IVIG at the beginning of the pandemic, when immunoglobulin was used as a therapeutic attempt for a then-unknown disease.

Therefore, the availability of new products, like V-IMMUNE produced by Virchow Laboratories in India, that are effective for the treatment of clearly defined indications and possess the necessary safety profile-ensuring minimal adverse reactions during and after clinical use-is essential.

The investigators present here a clinical trial for regulatory approval of a novel immunogloblin V-IMMUNE® in the Brazilian market for primary immunodeficiency.

Objectives

The objectives of the study are:

1. To evaluate the efficacy of the human normal immunoglobulin preparation V-IMMUNE® for patients with primary humoral immunodeficiency in preventing the rate of serious bacterial infection in 12 months compared to historical controls;
2. To evaluate the safety of the human normal immunoglobulin preparation V-IMMUNE® regarding the observed proportion of infusions with one or more temporally associated adverse events in patients with primary humoral immunodeficiency;
3. To evaluate the pharmacokinetics of intravenous V-IMMUNE® in patients with primary humoral immunodeficiency.

   Methods:

   Study Design This is a prospective, Phase III, open-label, non-randomized, multicenter, single-group study with a historical control for the regular administration of V-IMMUNE® via the intravenous route.

   Recruitment Plan Recruitment will take place through 10 national reference immunology centers specialized in the treatment of primary immunodeficiency with intravenous immunoglobulin infusion. Patients who are already receiving regular intravenous immunoglobulin therapy and meet the eligibility criteria will be invited to participate in the study, switching from their current product to the investigational product (IP) for a duration of 12 months.

   Recruitment Approach Patients who meet the inclusion criteria and are already receiving IgG treatment at the participating centers will be approached for inclusion in the VIP study. Once the informed consent form (ICF) is signed, the participant will begin receiving V-Immune® (On-Pharma) as per the study protocol.

   As this is a single-group study, randomization will not be performed. Blinding Given that this is a single-group study and the eligible patients are already being treated with another commercially available immunoglobulin, which will be replaced by V-IMMUNE®, blinding is deemed unnecessary.

   Experimental Intervention The Investigational Product (IP) is V-IMMUNE®, normal human immunoglobulin I.P. 5% (5g/100 mL), manufactured from qualified human plasma for intravenous use. Each vial contains Human Immunoglobulin 50 g/L, Maltose 100 g/L, and Water for Injection. The 5% Human Immunoglobulin solution for intravenous administration I.P. is a sterile, pyrogen-free preparation of normal human immunoglobulin in a single-dose form for intravenous infusion. Each 10 mL, 50 mL, and 100 mL contains 0.5 g, 2.5 g, and 5 g of normal human immunoglobulin, respectively, and is prepared from qualified human plasma using membrane filtration, combined chromatographic steps, and viral inactivation procedures. The IgA content does not exceed 2 mg/mL. The IgG subclass distribution is similar to that found in normal human serum.

   The manufacturing process uses plasma collected from donors who are screened based on medical history, in accordance with regulatory authority guidelines. The blood is tested for mandatory infectious diseases. Only plasma that tests negative for HBsAg, HCV, and HIV antibodies is used in the process.

   Normal Human Immunoglobulin I.P. 5% (5g/100 mL) V-IMMUNE® will be administered at a dose of 600 mg/kg every 3 weeks (+/- 3 days) via intravenous (IV) route at the infusion rate specified below, over a duration of 3 to 6 hours:

   0.01 ml/kg/min 0-30 min, 0.02 ml/kg/min 31 to 45 min, 0.04 ml/kg/min 46 to 60 min and 0.06 ml/kg/min 61 min until the end of infusion.

   Dose Escalation Dose escalation occurs gradually unless adverse events (AEs) occur. The dose is only increased if there is good tolerance, without the presence of adverse events. If an AE occurs, the infusion must be paused for 20 to 30 minutes. The use of loratadine, paracetamol, and ondansetron will be allowed. Exceptionally, another drug from the same class may be used, provided the pharmacokinetics study center is informed. Once the patient improves, the infusion is resumed at a reduced rate, returning to the initial infusion speed. The patient will be observed for 60 minutes after the infusion ends for clinical assessment and monitoring of potential adverse events .

   Pre-medication Pre-medication prior to infusion of the investigational product: rapid infusion of 500 mL of 0.9% sodium chloride (NaCl) IV, diphenhydramine 50 mg IV, and hydrocortisone 200 mg IV, followed by the investigational product administered at progressively increasing infusion rates as described above. After infusion, 0.9% NaCl should be continued at 1 mL/kg/hour. The use of pre-medication is standard medical practice and is considered necessary for participant safety.

   Rapid isotonic saline infusion before administration and slow isotonic saline infusion to maintain venous access for at least 30 to 40 minutes are necessary and standard practice in the administration of these blood products. Rapid crystalloid before infusion reduces the risk of headaches and aseptic meningitis post-administration, as well as the risk of thromboembolic events. Crystalloid administration after the investigational product infusion reduces the risk of serious and potentially life-threatening adverse events due to anaphylactic reactions by allowing for the rapid administration of IV medications in a potentially shocked patient, avoiding the need for emergency central venous access.

   Pre-medication Summary:

   Rapid infusion of 500 mL of 0.9% sodium chloride (NaCl) IV

   Diphenhydramine* 50 mg IV (adult); Pediatric: 1.25 mg/kg IV

   Hydrocortisone** 200 mg IV (adult); Pediatric: 3 mg/kg IV

   After infusion: 0.9% NaCl at 1 mL/kg/hour for one hour After the initial three months, diphenhydramine and hydrocortisone may be discontinued.

   Thromboembolism risk: use the slowest possible infusion rate

   * Administer 30 minutes before infusion.

   ** Administer 30 minutes to 1 hour before infusion.

   For individuals at risk of thromboembolism, the infusion rate must be kept as low as possible.

   Thromboembolism risk factors include: advanced age, obesity, hypertension, diabetes mellitus, history of previous thromboembolic events, known acquired or congenital thrombophilic disorders, prolonged immobilization, severe hypovolemia, or increased blood viscosity.

   Treatment intervals between administrations should remain constant throughout the study, provided that the IgG trough levels remain >500 mg/L.

   If body weight changes by more than 5% compared to baseline (screening visit), the dose will be adjusted to maintain a consistent mg/kg body weight dosage.

   In the event of clinically significant hypotension and/or anaphylactic reactions, in addition to stopping the infusion and administering appropriate supportive care (which may include epinephrine, antihistamines, corticosteroids, supplemental oxygen, and volume expansion), and recording the incident in the CRF as an AE, the participant may be withdrawn from the study at the investigator's discretion. In such cases, participants may, if they wish, complete follow-up visits

   Contraindications and Precautions Related to the IP Normal Human Immunoglobulin for Intravenous Administration I.P. 5% is contraindicated in patients with selective IgA deficiency.

   Patients may experience severe hypersensitivity reactions or anaphylaxis in the presence of detectable IgA levels after infusion of Normal Human Immunoglobulin I.P. 5%. The occurrence of severe hypersensitivity reactions or anaphylaxis under such conditions should prompt consideration of alternative therapy.

   The intravenous solution of Normal Human Immunoglobulin should only be administered intravenously.

   Additional listed precautions regarding the use of Normal Human Immunoglobulin I.P. 5% include:

   Hypersensitivity: Immediate hypersensitivity and anaphylactic reactions are rare but possible. If hypersensitivity occurs, immediately stop the infusion and initiate appropriate treatment. Medications such as epinephrine and antihistamines should be readily available for the immediate treatment of acute hypersensitivity reactions, including anaphylaxis.

   Renal dysfunction: Acute renal failure, osmotic nephropathy, and death may occur with IVIG use. Ensure that the patient is not hypovolemic prior to administration. In patients at risk of renal dysfunction due to pre-existing renal insufficiency or predisposition to acute renal failure (e.g., diabetes mellitus, hypovolemia, obesity, use of nephrotoxic medications, or age >65), IVIG should be administered at the minimum infusion rate.

   Aseptic Meningitis Syndrome (AMS): Rarely occurs with IVIG treatment. May begin within hours to 2 days after treatment. Discontinuation of IVIG usually leads to full recovery without sequelae. More common with high doses (2 g/kg) and/or rapid infusion.

   Hemolysis: IVIG products may contain blood group antibodies that act as hemolysins, coating red blood cells and causing a positive direct antiglobulin test and, rarely, hemolysis. Delayed hemolytic anemia may occur due to red cell sequestration and acute hemolysis, consistent with intravascular hemolysis.

   Transfusion-Related Acute Lung Injury (TRALI): Non-cardiogenic pulmonary edema may occur after IVIG administration. TRALI is characterized by severe respiratory distress, pulmonary edema, hypoxemia, normal left ventricular function, and fever, typically occurring 1 to 6 hours post-treatment. Patients should be monitored for pulmonary adverse events. If TRALI is suspected, appropriate tests should be conducted for anti-neutrophil antibodies in both the product and patient serum. Treatment includes oxygen therapy and ventilatory support.

   Transmissible Agents: Normal Human Immunoglobulin I.P. 5% is derived from human plasma. Due to effective donor screening and manufacturing processes, the risk of viral disease transmission is extremely low. The theoretical risk of Creutzfeldt-Jakob disease (CJD) transmission is also considered extremely remote.

   Monitoring - Laboratory Tests: Periodic monitoring of renal function and urine output is crucial in patients at increased risk of acute renal failure. Renal function (including serum urea and creatinine levels) should be assessed before the initial infusion and periodically as per the visit schedule. Due to a potentially increased risk of thrombosis, baseline blood viscosity assessment should be considered in patients at risk of hyperviscosity, including those with cryoglobulinemia, fasting chylomicronemia/markedly elevated triglycerides, or monoclonal gammopathies. If signs/symptoms of hemolysis are observed post-infusion, appropriate lab tests should be conducted. In cases of suspected TRALI, tests for anti-neutrophil antibodies should be performed on the product and patient serum.

   Patient Information: Patients should be instructed to immediately report symptoms such as decreased urine output, sudden weight gain, fluid retention, edema, and/or shortness of breath-which may indicate kidney injury.

   Pregnancy - Category C: Reproduction studies in animals have not been conducted with Normal Human Immunoglobulin for IV use. It is also unknown whether it can cause fetal harm when administered to a pregnant woman or affect reproductive capacity. It should be used during pregnancy only if absolutely necessary. Pregnant women are part of this study's exclusion criteria.

   Presentation of the Investigational Product (IP) Normal human immunoglobulin for intravenous administration I.P. 5%, V-IMMUNE®, is available in vials of 0.5g/10 mL, 2.5g/50 mL, and 5g/100 mL (5% concentration), in single-dose format for intravenous administration.

   IP Manufacturing and Labeling V-IMMUNE® immunoglobulin is manufactured, packaged, and labeled by Virchow Biotech Private Limited, and imported by OnPharma Importadora Exportadora e Distribuidora de Medicamentos LTDA, in accordance with current regulations. The preparation and labeling of the IP follow Good Manufacturing Practice (GMP) guidelines, and its distribution adheres to Good Distribution Practice (GDP) guidelines. IP labels will be in Portuguese and meet Brazilian legal requirements.

   Storage and Use Conditions of the IP V-IMMUNE® immunoglobulin must be stored in a secure area with limited access, preferably in a locked cabinet, protected from light, and kept at a temperature between 2°C and 8°C. V-IMMUNE® must not be frozen.

   Patient Confinement Procedures Patients not selected for pharmacokinetic (PK) analysis must arrive at the study centers 60 minutes before infusion and remain under observation for 60 minutes after the infusion ends for clinical assessment and monitoring for adverse events.

   For patients selected/eligible for PK analysis, the same confinement period will apply on infusion days 1 to 8 and 10 to 17. However, on day 9, these patients must arrive 60 minutes before the infusion and remain at the center for up to 6 hours after the infusion for blood sample collection. They must also return for blood draws at 24 hours, 72 hours, 7 days, 14 days, and 21 days after the 9th infusion.

   Pharmacokinetic Parameters

   The following pharmacokinetic parameters will be determined for this study:

   Cmax: Maximum plasma concentration reached, based on experimental data obtained directly from the plasma concentration-time curve.

   AUC₀-t (Area Under the Curve): Area under the plasma concentration-time curve from time zero to the last concentration above the lower limit of quantification, calculated using the trapezoidal rule.

   AUCinf: Area under the plasma concentration-time curve from time zero to infinity (extrapolated), calculated as AUCinf = AUC₀-t + Ct/Kel, where Ct is the last measurable concentration and Kel is the elimination rate constant.

   Tmax: Time to reach Cmax. Kel: Elimination rate constant, estimated from the slope of the linear regression of the natural logarithm of concentration versus time for at least three data points above the lower limit of quantification.

   T½ (Half-life): Elimination half-life, calculated as ln(2)/Kel. Vd (Volume of distribution): Volume of distribution from the terminal phase of the pharmacokinetic curve, calculated as Dose/(Kel × AUCinf).

   Sampling Schedule Samples will be collected using 7.5 mL tubes with gel separators, labeled with participant number, collection number, timepoint, infusion number, product code (IGG), and protocol number. Blood samples of 7.5 mL each will be collected before infusion number 0 (prior IVIG treatment used by the participant) and before infusions 1 to 9 of V-IMMUNE®.Post-infusion pharmacokinetic samples will be collected following the ninth (9th) infusion Analytical Stage According to the literature, the analytical phase involves a sample preparation method based on enzymatic digestion with trypsin. This may be preceded by reduction and/or alkylation followed by enzymatic digestion.

   The cited preparation approach aims to develop and apply a robust and selective MRM (Multiple Reaction Monitoring) method, capable of detecting a specific Q1/Q3 ion pair derived from the digestion of the target protein-in this case, IgG-thus indirectly determining its plasma concentration. Given the existence of 4 IgG subclasses (IgG1, IgG2, IgG3, and IgG4), specific peptide fragments can be found in protein databases and scientific literature that are unique to each subclass. The following peptide sequences have been adopted as the starting point for the development of the bioanalytical method for quantifying total IgG and its subclasses:

   Peptide FNWYVDGVEVHNAK - specific for IgG1 Peptide CCVECPPCPAPPVAGPSVFLFPPKPK - specific for IgG2 Peptide WYVDGVEVHNAK - specific for IgG3 Peptide TTPPVLDSDGSFFLYSR - specific for IgG4 Since the analyte is an endogenous substance, a bioanalytical method using a surrogate matrix (in this case, bovine plasma) is necessary. This surrogate will be used to generate calibration curves and quality control samples processed in a similar manner to the unknown samples from study participants.

   For sample preparation and LC-MS/MS analysis, the following reagents may be used if extraction with prior reduction and alkylation is required: ammonium bicarbonate, 2,2,2-trifluoroethanol, DL-dithiothreitol, iodoacetamide, formic acid or acetic acid, among others. If only protein precipitation followed by enzymatic digestion is performed, reagents such as acetone, isopropanol, perchloric acid, acetonitrile, or methanol may be used.

   In both cases, the sample must be incubated with MS-grade trypsin at a minimum suggested concentration of 1 g/L.

   Chromatographic methods will employ mobile phase gradients to improve separation of the various peptide chains that may be formed during extraction. The system will operate at pressures compatible with UPLC, with an aqueous mobile phase containing 0.1% formic acid and an organic phase consisting of methanol or acetonitrile, also with 0.1% formic acid. Recommended columns include solid-core types such as Waters X-Bridge C8 (3.0 × 30 mm, 3.5 µm) or Agilent Eclipse Plus C18 RRHD (1.8 μm, 2.1 × 100 mm).

   Detection of the analytes will be performed using a triple quadrupole mass spectrometer, model API6500 from Sciex. The method will be validated in accordance with RDC No. 27, dated May 17, 2012, covering the validation parameters of linearity, precision, accuracy, carryover, matrix effect, selectivity, stability in biological matrix, and solution stability Control or Standard Treatment: The control group will consist of historical controls as described in the literature Co-interventions: No co-interventions will be allowed. Follow-up For 12 months.

   Visits:

   • All immunoglobulin infusion opportunities with data collection - it is anticipated that there will be 17 visits for V-IMMUNE® infusion during 1 year. Patients will be observed:
   * Immediately before infusion;
   * During infusion and up to 60 minutes after;
   * 24 and 72 hours after the start of infusion of the investigational product - by telephone contact.

   Laboratory data:

   At "Baseline", and before performing 1st, 3rd, 6th, 9th, 12th, and 17th infusions:

1. BHCg, CBC, platelets, electrolytes, serum glucose, urea, creatinine, AST, ALT, LDH, total and partial urine bilirubin (type 1)

Before performing 1st, 3rd, 6th, 9th, 12th, and 17th infusions:

1. Haptoglobin, Coombs

Before all infusions:

1. Trough IgG Screening Visits (T1 and T2)

Objective:

Identify eligible patients by evaluating inclusion and exclusion criteria, measuring IgG levels, and obtaining informed consent.

Activities at Screening Visit T1: Reception and Informed Consent:

Provide a detailed explanation of the study, including objectives, procedures, risks, and benefits.Written informed consent (ICF/Assent) must be obtained by qualified and delegated personnel and signed by the investigator before any study procedures or screening labs are conducted.

Assess time since primary immunodeficiency diagnosis. Assess premedication use with prior IgG infusion. Check osmolarity and IgA content of previous IgG which was in use. Assess adherence to previous IgG treatment schedule (infusion frequency and two most recent trough levels).

Obtain written informed consent.

Demographic and Medical History Data Collection:

Record age, sex, race, weight, and BMI. Collect medical history, including infections and current medications.

Eligibility Criteria Assessment:

Review inclusion criteria (e.g., confirmed diagnosis, appropriate age). Evaluate exclusion criteria (e.g., autoimmune disease, IgG allergy to previous IgG brand in use).

Physical and Clinical Examination:

Perform a physical exam. Record vital signs (RR, HR, BP, temperature).

Sample Collection for Lab Tests:

Baseline IgG levels:

If two prior IgG levels >500 mg/dL within 90 days, patient may proceed without new screening lab.

If one prior IgG level >500 mg/dL within 30 days, proceed to T2 for second test.

If IgG at T1 >700 mg/dL within 30 days, infusion may proceed at T2 even before T2 result.

Other labs per protocol. Quality of Life and Symptom Questionnaires:Apply SF-36 QoL questionnaire. Assess current symptoms related to the condition.

Activities at Screening Visit T2:

Reassess IgG treatment adherence. echeck inclusion/exclusion criteria. Repeat physical exam and vitals. Collect second IgG sample if needed (may occur same day as first infusion if prior level >700 mg/dL).

Other protocol-specific labs. Flexible window: Screening can be extended (investigator's discretion) until baseline IgG >500 mg/dL is confirmed.

First Infusion Visit (I1) Objective: Confirm eligibility and start IP administration.

Activities:Review Screening Results:

Review lab findings and eligibility criteria. Discuss abnormal results and eligibility status.

Clinical Assessment:

Update physical exam and vital signs. Review health status changes. Provide symptom diary instructions.

Eligibility Confirmation:

Final eligibility confirmation. Review concomitant medications.

Lab Sample Collection:

Baseline IgG. Pregnancy test for women of childbearing age unless permanently sterile. Other tests: CBC with platelets, electrolytes, glucose, urea, creatinine, AST, ALT, LDH, urinalysis, pneumococcal and Haemophilus antibody titers.

Pre-dose IgG from prior product. Pre-dose PK samples.

First Infusion of V-Immune®:

Explain procedure. Record batch number and expiration date. Administer per infusion protocol.

Monitor for adverse events (AEs):

Record AE, infusion rate at onset, interruptions, restart rate, total infusion time, total IgG dose, and premedication use.

Antibodies anti-polissacaride for pneumococcus and Haemophylus

Post-Infusion Data Collection:

Record AEs, post-infusion vitals (30-60 min), and general condition. Record discharge time.

Patient Instructions:

Provide post-infusion guidance, emergency instructions, and team contact. Inform that follow-up calls will occur at 24 and 72 hours. Schedule next visit. Infusions 2 to 16 (I2 to I16) Objective: Conduct infusions every 3 weeks (±3 days).

Activities:

Review Previous Results and Clinical Status:

Review previous labs and symptoms. Update physical exam and vitals. Review infections, hospitalizations, antibiotics, time to resolution, and workdays lost.

SF-36 at infusions 8 and 16 for adolescents and adults. AUQEI will be used for children

Lab Collection:

Pre-infusion IgG for all visits. Pre-dose PK samples for infusions 1-9. Pos-dose will be 16 PK samples per adult ; children only pre-dose. (9 samples) Infuions 3, 6, 9, 12, 17: pregnancy test for women of childbearing potential. Other labs: CBC, electrolytes, glucose, urea, creatinine, AST, ALT, LDH, urinalysis, haptoglobin, Coombs test.

*Infusion 6: pneumococcal and Haemophilus antibody titers.

V-Immune® Infusion:

Record batch and expiration. Administer per protocol. Monitor and document AEs and all infusion details.

Post-Infusion:

Record AEs, post-infusion vitals (30-60 min), discharge time, PK per section

Patient Instructions:

Post-infusion guidance, team contact, 24h/72h follow-up calls, next visit scheduling.

Physical Examination

Conducted by qualified staff, includes:

General appearance, head/ENT, thorax, cardiovascular, respiratory, abdomen, musculoskeletal, genitourinary, skin.

Clinically significant changes are recorded as AEs. Vital Signs

To be consistently collected in the same position:

Systolic/diastolic BP, HR (bpm), RR (breaths/min), temperature (°C). Final Infusion and End-of-Study Visit

Activities:

Severe Infections per Patient-Year:

Total number, type, treatment, and outcomes.

Infusions with AEs:

Total infusions vs. number with AEs.

Safety and AE Assessment:

Infusion-related AEs: severity, duration, outcome, causality. Serious AEs (SAEs): details, actions, outcomes.

Overall Clinical Assessment:

Complete physical exam, vital signs.

Quality of Life:

SF-36, patient satisfaction.

Treatment Adherence:

Confirm monthly infusions, missed/delayed doses, reasons.

Final Participant Debriefing:

Summary of treatment, post-study follow-up plans.

Final Visit Procedures:

Check-in, contact updates, document AEs, discuss outcomes and study closure. Strategies to Minimize Loss to Follow-Up Missed Visits and Scheduled Sample Deviations Reschedule within 7 days. Mark as "missed/unavailable" if patient cannot attend.Only classified as loss to follow-up if no contact is possible by study end despite all efforts.

Patient Withdrawal from the Study

Occurs if:

Requested by patient. Two consecutive or three total missed visits. Development of HBV, HCV, or HIV. SAE making further IP dosing inappropriate (investigator discretion). Use of exclusionary medications Withdrawal of Consent A participant will be considered to have "Withdrawn Consent" if they choose to discontinue participation in any further study procedures. This right will be acknowledged and confirmed through the Informed Consent Form (ICF/Assent Form). Once consent is withdrawn, no additional study procedures will be carried out and no further data will be collected. Data collected up to the point of withdrawal will remain in the study database; however, if the participant requests the removal of their data, it will not be used.

Sample size calculation and statistical analysis plan. The investigators will include 50 patients to meet the sample size required to evaluate efficacy

Safety:

41 participants with at least complete data provides with a 90% probability of finding an upper limit of the one-sided 95% confidence interval < 0.40, assuming that the true observed proportion of infusions with one or more temporally associated AE is less than 20%. National data corroborate the above premise

Efficacy:

50 participants are required. Assuming a serious infection rate per person-year < 1, the investigators will have a 90% power to reject the one-sided H0 that the serious infection rate ≥ 1 per person-year, with a 1% significance level and 20% loss to follow-up. This number is compatible with the FDA rule that suggests that the upper limit of the 99% confidence interval should be < 1 serious infection per person-year. The investigators plan an interim analysis after 6 months of treatment or when 50% of the sample is reached, whichever occurs first, with a significance level of 0.5%, based on the Pocock criterion , to maintain an overall significance level of 1%.

Pharmacokinetics:

Number of patients per age group follows EMA recommendations. There will be 20 participants adult and adolescent participants aged 16 years or older, 6 children from 2 to 12 yo and 6 children from 13 to 16 yo. As recommended by the EMA, trough values will be collected for children, but without a complete pharmacokinetic curve in order to reduce the burden of multiple blood collections for this age group. Participants are the same as those in the efficacy and safety study.

Antibody measurement 3.9.1 Measurement parameters

For the present study, the following antibodies will be measured:

Anti-pneumococcal capsular polysaccharide Anti-Haemophilus influenzae: Assessment of antibodies against Haemophilus influenzae type b allows evaluation of the competence of the humoral immune response against encapsulated antigens.

It is a relevant parameter for identifying defects in antibody production, commonly used in the investigation of primary immunodeficiencies.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 2 years or older;
* Primary immunoglobulin G deficiency, already receiving another intravenous immunoglobulin (IVIG). Primary IgG deficiency may be secondary (non-exhaustive list) to one of the following diagnoses:
* Agammaglobulinemia due to absence of B cells
* Hypogammaglobulinemia with reduced antibody function - variable common immunodeficiency complex
* Quantitative and functional deficiencies of immunoglobulin G
* Normal immunoglobulin with reduced capacity for antibody production after immunization (e.g., Wiskott-Aldrich syndrome, IgG subclass deficiency, antipolysaccharide antibody deficiency against Haemophilus or pneumococcus)
* Severe combined immunodeficiencies: DiGeorge syndrome presenting with immunoglobulin G deficiency
* Isotype-switching defects: hyperimmunoglobulinemia M syndromes
* Two trough IgG measurements ≥500 mg/dL within the past 90 days.
* Participants with through IgG measurements ≥700 mg/dL within the last 30 days before the first visit

Exclusion Criteria:

* Acute infection under treatment within 2 weeks prior to screening
* Pregnancy
* History of hypersensitivity reaction to blood or blood products
* Previous anaphylactic reaction to IgG
* Intolerance to any component of V-Immune
* IgA deficiency, history of reactions to products containing IgA, or history of anti-IgA antibodies
* Selective Deficiency of IgA, IgM, IgD, or IgE
* Participation in any other study involving an investigational product
* Exposure to blood or any blood-derived products in the last 3 months
* Known HIV, HCV, or HBV infection
* ALT >3× the upper limit of normal or 3x baseline value
* Serum creatinine >2× the upper limit of normal or 2x baselline value
* BUN >2.5× the upper limit of normal or 2.5x baseline value
* History of NYHA class III/IV heart failure
* Uncontrolled hypertension with systolic BP >160 mmHg or diastolic BP >100 mmHg
* History of thrombotic events such as DVT, MI, stroke, or PE within the last 6 months
* Neoplasia under treatment
* Severe hepatic, renal, or cardiac insufficiency
* Child-Pugh class B/C hepatic insufficiency
* Alcohol, opioid, or psychotropic drug abuse within the last 12 months
* Use of immunosuppressive agents
* Long-term use of prednisone >10 mg/day or equivalent
* Protein-losing enteropathies (Crohn's disease, ulcerative colitis, Ménétrier's disease, celiac disease)

Observation:

If Research participant becomes pregnant during study participation - we will Discontinue any further administration of the IMP; The principal investigator must refer the research participant for follow-up through routine healthcare services; The research participant will continue to be monitored by the study; Obtain informed consent from the pregnant participant to request authorization to follow her pregnancy; If authorized by a specific informed consent form, even after the participant's involvement in the study has ended, the investigator must contact the pregnant participant quarterly to monitor the pregnancy. The results of this follow-up must be entered into the CRF. The frequency will be maintained as long as no abnormalities are identified in the participant, the pregnancy, or the fetus.

Female partner of a male research participant becomes pregnant during the study = No action is required regarding the research participant's participation; Obtain informed consent from the research participant's partner to request authorization to monitor her pregnancy. If authorized by a specific informed consent form, the investigator must contact the pregnant woman quarterly to monitor the pregnancy. The results of this follow-up must be entered into the CRF. The frequency will be maintained as long as no abnormalities are identified in the pregnant woman, the pregnancy, or the fetus.

Data Confidentiality:

The confidentiality of data from all patients will be ensured and preserved. Patient identification will be performed exclusively through the study-assigned identification number, the patient's initials, and date of birth. An exception to this procedure applies to participants included in the pharmacokinetic analyses, who, after providing consent themselves or through their legal representative, will also have their personal identifying data (full name, CPF [Brazilian individual taxpayer registry number], date of birth, and sex), as well as information regarding their participation (date of study enrollment), collected and transferred to the ICF laboratory for registration in the SINEB system (Sistema de Informações de Estudos de Equivalência Farmacêutica e Bioequivalência), an ANVISA database used for the registration of participants in studies of this nature.

Data obtained from medical records and other documents will be maintained in a confidential manner by the research centers and stored in locations with restricted access limited to the study team. Sensitive data, such as patient contact information collected for scheduling and follow-up purposes, will be accessed exclusively by personnel involved in the conduct of the study. The principal investigator shall allow direct access to participants' records and source documents for the purposes of monitoring, auditing, or inspection by the Sponsor and Regulatory Authorities, if required.

With regard to participants included in the pharmacokinetic analyses, the collection of personal identifying data (full name, CPF [Brazilian individual taxpayer registry number], date of birth, and sex) and participation-related information (date of study enrollment) is planned for transfer to the ICF laboratory for registration in the SINEB database. This procedure aims to mitigate risks to research participants by ensuring that they are not concurrently enrolled in another study within an interval shorter than six (6) months.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-08-15 (Actual); Primary Completion 2026-09-27 (Estimated); Study Completion 2027-02-27 (Estimated)

PRIMARY OUTCOMES:
Efficacy primary outcome | 12 months
  The primary efficacy endpoint is the rate of serious bacterial infections per person-year. These serious bacterial infection are: bacteremia/sepsis, bacterial meningitis, osteomielitis/septic arthritis, bacterial pneumonia, visceral abscess Definition of each serious bacterial infection are stated accordinly in the protocol.
Safety outcome | 72 hours
  Proportion of infusions with one or more temporally associated adverse events (AEs)

SECONDARY OUTCOMES:
Severe and non-severe bacterial infections | 12 months
  Relationship of severe and non-severe bacterial infections to:
  The product dose
  Which infusion they occurred after (e.g., 1st, 2nd, 3rd, etc.)
  The nadir of total IgG levels
  Antibody levels against pneumococcal capsular polysaccharide and Haemophilus influenzae
Number of patients with 0, 1, 2, etc., severe infections | 12 months
  Proportion of patients with 0, 1, 2, etc., severe infections
Number of adverse events by body systems | 12 months
  Number of adverse events by cardiovascular, gastrointestinal, neurological, renal, hepatic, motor, and respiratory systems
Time to first infection | 12 months
  Time in days to first infection
Nadir of pre-infusion total IgG level | 3 weeks
  Value of pre-infusion total IgG level in adults prior to each infusion
Nadir of pre-infusion total IgG level in children aged 2 to <16 years | 3 weeks after the fifth infusion
  Value of pre-infusion total IgG level in children aged 2 to <16 years, starting from the fifth infusion
Number of any severe or non-severe infection | 12 months
  Total Number of any severe or non-severe infection (total and by category)
Infection resolution time | 12 months
  Time taken to severe infection resolution
Use of antibiotics | 12 months
  Number of antibiotics (antibiotic treatment) use per patient
Hospitalizations due to infections | 12 months
  Number of Hospitalizations due to infections
Episodes of fever | 12 months
  Number of Episodes of fever per patient
Number of days absent from school or work | 12 months
  Total Number of days absent from school or work due to infections and treatment
Quality of life: Short Form Health Survey (36) | 6 and 12 months
  Questionnaire of quality of life SF-36 at 6 and 12 months for adolescents and adults.The 8 Domains of the SF-36: Physical Functioning, Role Limitations due to Physical Health, Bodily Pain, General Health Perceptions, Vitality, Social Functioning, Role Limitations due to Emotional Problems and Mental Health Measures general mental health, including depression and anxiety. Scoring: Each domain is scored separately from 0 to 100 0 = worst health 100 = best health Scores are calculated using a weighted algorithm specific to the questionnaire. Items are coded, summed, and transformed into a scale from 0-100 according to the scoring manual.
Minimum total IgG level (500 mg/dL) not reached | 12 months
  Proportion of individuals who did not reach the target minimum total IgG level (500 mg/dL) at any time on or after five estimated half-lives
Trough total IgG measurement | 12 months
  Trough total IgG measurement for each infection
Secondary safety outcome | 12 months
  The total number of AE that occur during or within 72 hours of an infusion
Secondary safety outcome | 12 months
  Average number of temporally associated AEs (within 72 hours of an infusion) per infusion, calculated as the ratio of (i) ÷ (ii):
  i. the total number of AEs that occur during or within 72 hours of an infusion ii. the total number of infusions
Secondary safety outcome | 12 months
  Proportion of patients who experienced one or more AEs at any time during the clinical study
Number of adverse events by cardiovascular, gastrointestinal, neurological, renal, hepatic, motor, and respiratory system assessed by CTCAE 4.0 | 12 months
  Count of the Number of events in each system (cardivoascular, gastrointestinal, neurological, renal, motor, hepatic and respiratory
Proportion of participants who could not reach minimum target level of Total Immunoglobulin ≥ 500 mg/dL | 5 estimated half-lives
  Percentage of participants who could not reach minimum target level of Total Immunoglobulin ≥ 500 mg/dL measured in any time equal or superior to 5 estimated half lives
Trough total IgG level per infection | at each occurrence of an infection.
  Dosage of Trough total IgG level in each infection

OTHER OUTCOMES:
Cmax | 12 months
  Maximum plasma concentration achieved, based on experimental data, obtained directly from the plasma concentration versus time curve.
ASC0-t | 12 months
  Area under the plasma concentration versus time curve, from time 0 to the time of the last concentration observed above the lower limit of quantification (calculated using the trapezoidal method)
Tmax | 12 months
  Time at which Cmax occurs
Kel | 12 months
  Elimination rate constant, estimated from the slope of the regression line calculated by the least squares method using the natural logarithm of concentration versus time for the last values (at least three) above the lower limit of quantification
T1/2 | 12 months
  Half life of elimination, calculated as ln(2)/Kel
Vd | 12 months
  Volume of distribution obtained from the terminal phase of the pharmacokinetic curve, calculated as Dose / (Kel × AUCinf)

CONTACTS AND LOCATIONS:
Overall Officials: Israel Silva Maia, PhD, Study Chair — Hospital do Coracao; Dewton Moraes Vasconcelos, PhD, Principal Investigator — Hospital do Coracao
Locations (1):
- IMIP Centro de Pesquisa, Recife, Pernanbuco, Brazil

IPD SHARING:
Plan to Share IPD: No
Due to the regulatory nature of this clinical trial-specifically aimed at obtaining market authorization for V-IMMUNE® in Brazil for patients with immune thrombocytopenia-we will not be able to share individual participant data (IPD) outside of the study team. All participant information is considered proprietary and confidential as part of the registration dossier being submitted to the Brazilian health authority. The study protocol, data collection, and analyses must remain under restricted access to fulfill legal, regulatory, and institutional requirements, which include protecting patient privacy and maintaining data integrity for the product's approval process. Consequently, no external IPD sharing is planned at this time.

REFERENCES:
- [Background] FDA. 2008. Guidance for Industry: Safety, Efficacy, and Pharmacokinetic Studies to Support Marketing of Immune Globulin Intravenous (Human) as Replacement Therapy for Primary Humoral Immunodeficiency
- [Background] Goudouris ES, Silva AMDR, Ouricuri AL, Grumach AS, Condino-Neto A, Costa-Carvalho BT, Prando CCM, Kokron CM, Vasconcelos DM, Tavares FS, Segundo GRS, Barreto ICDP, Dorna MB, Barros MAMT, Forte WCN. Comment to: II Brazilian Consensus on the use of human immunoglobulin in patients with primary immunodeficiencies. einstein (Sao Paulo). 2017;15(1):1-16. Einstein (Sao Paulo). 2017 Oct-Dec;15(4):522. doi: 10.1590/S1679-45082017CE4250. No abstract available. PMID 29364371
- [Background] Buckley RH, Schiff RI. The use of intravenous immune globulin in immunodeficiency diseases. N Engl J Med. 1991 Jul 11;325(2):110-7. doi: 10.1056/NEJM199107113250207. No abstract available. PMID 2052044
- See also: Sponsor´s website — https://onpharma.com.br/